CLINICAL TRIAL: NCT03396757
Title: The Artificial Kidney Initiation in Kidney Injury 2 A Multi-Centre, Randomized, Controlled Trial
Brief Title: The Artificial Kidney Initiation in Kidney Injury 2
Acronym: AKIKI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K160916J; 2017-A02382-51 (Other: Sponsor code / IDRCB)
Record Dates: First submitted 2018-01-02; First posted 2018-01-11 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Renal Replacement Therapy for Acute Kidney Injury in ICU
Keywords: Acute Kidney Injury; Critical Care; Renal Replacement Therapy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard strategy (Active Comparator): RRT will be initiated within 12 hours after documentation of serum urea concentration >40 mmol/l and/or an oliguria/anuria for more than 72 hours (identical to the delayed strategy in AKIKI).
  Interventions: Procedure: Standard strategy
- Delayed strategy (Experimental): RRT will be considered only if one potentially severe following situation occurs (noticeable hyperkalemia, or acidosis or pulmonary edema due to fluid overload resulting in severe hypoxemia which do not respond rapidly to medical treatment) or if serum urea concentration reaches 50 mmol/L.
  Interventions: Procedure: Delayed strategy

INTERVENTIONS:
Procedure: Standard strategy — RRT is initiated within 12 hours after documentation of serum urea concentration >40 mmol/l and/or an oliguria/anuria for more than 72 hours. The timing of its initiation will be recorded and RRT will continue until criteria for cessation are observed. This arm corresponds to the "delayed strategy" in the published AKIKI trial (NEJM 2016),
  Arms: Standard strategy
Procedure: Delayed strategy — RRT will be initiated only if one or more of above-mentioned potentially severe situations occur (identical to those used during the observational study) or if serum urea concentration reaches 50 mmol/L (this level being chosen in order to avoid extreme elevations of serum urea levels as mentioned above). The physician in charge will be allowed to try a medical treatment. Patients will not receive RRT whatever the duration of anuria/oliguria if any above-mentioned indication for RRT is not present. When required, RRT will be performed with the same modalities and stopped according to the same criteria as in the "no further delayed" RRT strategy, with special care to avoid dialysis disequilibrium syndrome (see below).
  The decision to initiate RRT in the "delayed strategy" arm of the trial will have to be approved by the attending physician(s) involved in patient's care in order to make sure that it corresponds to her/his usual practice.
  Arms: Delayed strategy

SUMMARY:
The timing of renal replacement therapy (RRT) in the context of severe acute kidney injury (AKI) is one the most debated issues in critical care medicine. The Artificial Kidney Initiation in Kidney Injury (AKIKI) was the first large prospective multicenter randomized trial published on this topic. This study (published in the New England Journal of Medicine, July 2017) showed no significant difference between an early and delayed RRT initiation strategy in term of mortality. Nearly 50% of patients escaped RRT in the delayed strategy and this strategy was associated with less catheter-related infections and faster renal function recovery. Two (serum urea concentration >40 mmol/l and oliguria/anuria for more than 72 hours) of the 5 criteria which mandated RRT in the delayed strategy are still open to debate since they have never been shown to put patient at danger. To go further into our investigation of RRT criteria, the investigators designed a study that would compare the "delayed strategy" used in AKIKI that can now be considered as "standard" with another in which RRT is delayed for a longer period in the absence of a life-threatening complication (such as hyperkalemia or severe overload pulmonary edema).

DETAILED DESCRIPTION:
The timing of renal replacement therapy (RRT) in the context of severe acute kidney injury (AKI) is one the most debated issues in critical care medicine. The Artificial Kidney Initiation in Kidney Injury (AKIKI) was the first large prospective multicenter randomized trial published on this topic. This study conducted by our team (published in the New England Journal of Medicine, July 2017) showed no significant difference between an early and delayed RRT initiation strategy in term of mortality. Nearly 50% of patients escaped RRT in the delayed strategy and this strategy was associated with less catheter-related infections and faster renal function recovery. Two (serum urea concentration >40 mmol/l and oliguria/anuria for more than 72 hours) of the 5 criteria which mandated RRT in the delayed strategy are still open to debate since they have never been shown to put patient at danger. To go further into our investigation of RRT criteria,the investigators designed a study that would compare the "delayed strategy" used in AKIKI that can now be considered as "standard" with another in which RRT is delayed for a longer period in the absence of a potentially severe complication (such as hyperkalemia or severe overload pulmonary edema).

The AKIKI 2 study will be a prospective, multicenter, open-label, two-arm randomized trial.

The study will involve 2 stages (an observational stage and a randomization stage) At any time during these two stages, the occurrence of a potentially severe condition defined below will mandate strong consideration for immediate RRT initiation unless a medical treatment can very rapidly resolve the situation.

Criteria that mandate strong consideration for RRT initiation at any time during the 2 stages of the study

1. Serum potassium concentration >6 mmol/l
2. Serum potassium concentration >5.5 mmol/l persisting despite medical treatment
3. Arterial blood pH <7.15 in a context of pure metabolic acidosis (PaCO2 <35 mmHg) or in a context of mixed acidosis with a PaCO2 >50 mmHg without possibility of increasing alveolar ventilation
4. Acute pulmonary edema due to fluid overload despite diuretic therapy leading to severe hypoxemia requiring oxygen flow rate >5 l/min to maintain SpO2>95% (oxygen saturation) or FiO2>50% (inspired oxygen fraction) under invasive or non-invasive mechanical ventilation

   * Observational Stage: All patients receiving (or who have received for the present episode) intravenous catecholamines and/or invasive mechanical ventilation and presenting with AKI classification stage 3 of KDIGO classification [defined by at least one of the following criteria: serum creatinine concentration of more than 4 mg/dl (354 µmol/liter) or greater than 3 times the baseline creatinine level, anuria (urine output of 100 ml/day or less) for more than 12 hours, oliguria (urine output below 0.3 ml/kg/h or below 500 ml/day) for more than 24 hours] and who have no potentially severe condition mandating strong consideration for immediate RRT initiation as described above will be included in an observational study. Clinical and metabolic conditions will be closely monitored and RRT consideration will be mandatory if one or more of these conditions (see above) occurs.
   * Randomization stage: Patients presenting, either immediately after inclusion or during their follow-up in the observational study, one or both of following criteria: a serum urea concentration >40 mmol/l and/or an oliguria/anuria for more than 72 hours even in the absence of an above-mentioned potentially severe condition will be randomly allocated to one of the two study treatment arms. One arm is termed "standard strategy" (which was the delayed arm of AKIKI 1) and the other a "delayed RRT strategy".

"Standard strategy": RRT is initiated within 12 hours after documentation of serum urea concentration >40 mmol/l and/or an oliguria/anuria for more than 72 hours. The timing of initiation will be recorded and RRT sessions will be performed until criteria for cessation are observed (see below).

"Delayed strategy": RRT will be initiated only if one or more of above-mentioned potentially severe situations (see "Criteria that mandate strong consideration for RRT initiation at any time") occur (identical to those used during the observational study) or if serum urea concentration reaches 50 mmol/L (this level being chosen in order to avoid extreme elevations of serum urea levels as mentioned above). As already explained, the physician in charge will be allowed to try a medical treatment of hyperkalemia, acidosis or pulmonary edema and the decision to start RRT or not will be taken by him, according to his usual practice. The duration of anuria will not constitute a criterion per se for RRT initiation. When required, RRT will be performed with the same modalities and stopped according to the same criteria as in the standard strategy, with special care to avoid dialysis disequilibrium syndrome.

The choice of RRT modality (intermittent or continuous technique) will be left at the study site discretion. Several RRT modalities can be used in the same patient, according to attending physician's indication. Duration of and interval between sessions, and device settings as well as modality of anticoagulation are left at the investigator's discretion. However, RRT will be prescribed and monitored according to national guidelines in order to ensure optimal efficacy of RRT.

In case of RRT initiation in a context of high serum urea concentration (> 40 mmol/l), prevention of dialysis disequilibrium syndrome will be recommended. The management will be left at clinician's discretion and will include one or several of the following measures :

* Slow, gentle initial hemodialysis (dialysis time <2 hours and low blood flow rate)
* Increasing dialysate sodium levels
* Administration of osmotically active substance by using a high-glucose-concentration dialysate or administering hypertonic glucose in the venous line of the dialyser during dialysis.

All study centers have extensive experience in both acute kidney injury management and RRT techniques.

Renal replacement therapy discontinuation will be contemplated when spontaneous diuresis >500 ml/24h, and highly recommended if diuresis is >1000 ml/24h without diuretic administration or >2000 ml/24h, in patients receiving diuretics.

Renal replacement therapy cessation will be mandatory if diuresis (as defined above) is present and serum creatinine level decreases spontaneously.

If improvement of renal function is insufficient to achieve a spontaneous decrease in creatinine level and/or if diuresis becomes lower than 1000 ml/24h without diuretics (or lower than 2000 ml/24h under diuretics), RRT will be resumed.

Renal function recovery will be defined according to urine output as mentioned above and RRT cessation without need for resumption in the following 7 days.

RRT will be initiated only if one or more of above-mentioned potentially severe situations occur (identical to those used during the observational study. The physician in charge will be allowed to try a medical treatment.) or if serum urea concentration reaches 50 mmol/L (this level being chosen in order to avoid extreme elevations of serum urea levels as mentioned above). Patients will not receive RRT whatever the duration of anuria/oliguria if none of the above-mentioned indications for RRT is present. When required, RRT will be performed with the same modalities and stopped according to the same criteria as in the "standard" RRT strategy, with special care to avoid dialysis disequilibrium syndrome.

The decision to initiate RRT in the "delayed strategy" arm of the trial will have to be approved by the attending physician(s) involved in patient's care in order to make sure that it corresponds to her/his usual practice.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be fulfilled to be included in the observational study (first stage):

* Adults (>18 years)
* Hospitalized in a study ICU.
* Evidence of acute kidney injury compatible with the diagnosis of acute tubular necrosis in a context of ischemic or toxic aggression and who receive (or received for the same episode) invasive mechanical ventilation and/or catecholamine infusion.
* Acute kidney injury stage 3 of KDIGO classification defined by at least one of the following criteria: serum creatinine concentration of more than 4 mg/dl (354 µmol/liter) or greater than 3 times the baseline creatinine level, anuria (urine output of 100 ml/day or less) for more than 12 hours, oliguria (urine output below 0.3 ml/kg/h or below 500 ml/day) for more than 24 hours.

To be randomized (randomization stage), supplemental criteria must be fulfilled. These criteria can appear either immediately after inclusion in the observational stage, or during the follow-up of the patient in the observational stage, in the absence of any non-inclusion criteria (listed below) at the time of randomization:

* Oliguria/anuria (urine output <0.3 ml/kg/h or <500 ml/day) for more than 72 hours or serum urea concentration comprised between 40 and 50 mmol/l.
* Affiliation to a social security regime

Exclusion Criteria:

* Severity criteria mandating immediate RRT initiation (Table 1)
* Serum urea level > 50 mmol/l
* Severe chronic renal failure (defined by a creatinine clearance < 30 ml/min)
* Patients with inclusion criteria already present for more than 24 hours (to avoid delayed inclusions)
* AKI caused by urinary tract obstruction or renal vessel obstruction or tumour lysis syndrome or thrombotic microangiopathy or acute glomerulopathy
* Poisoning by a dialyzable agent
* Child C liver cirrhosis
* Cardiac arrest without awakening
* Moribund state (patient likely to die within 24h)
* Patient having already received RRT for the current episode of AKI
* Renal transplant
* Treatment limitation (withholding or withdrawal)
* Previous inclusion in this study
* Subject deprived of freedom, subject under a legal protective measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
number of RRT-free days | Day 28 after randomization
  One point will be given for each calendar day during the measurement period (i.e. from the first day of randomization to day 28) that a patient was both alive and free of RRT, assuming the patient survives and remains free of RRT for at least 3 consecutive calendar days after RRT weaning, whatever the vital status at day 28. Zero value will be given for patients with RRT initiated the first day of randomization who died before RRT weaning or who remained under RRT until day 28.
  With this definition, RRT-free days may concern days without RRT both before RRT initiation (a situation encountered by definition in the " delayed strategy" arm) and after RRT weaning (for the two strategies).

SECONDARY OUTCOMES:
Hydration status (randomization stage) | Until ICU discharge or day 28 after randomization
  weight
Hydration status (randomization stage) | Until ICU discharge or day 28 after randomization
  clinical edema scale
Hydration status (randomization stage) | Until ICU discharge or day 28 after randomization
  fluid balance
Nutritional status (randomization stage) | Until ICU discharge or day 28 after randomization
  Amount of calories and protein administered
Nutritional status (randomization stage) | Until ICU discharge or day 28 after randomization
  serum albumin, transthyretin and CRP (C Reactive Protein) concentration changes
Number of hemorrhages (randomization stage) | Until ICU discharge or day 28 after randomization
  hemorrhages requiring red blood cell transfusion or surgical procedure
Rate of thrombocytopenia (randomization stage) | Until ICU discharge or day 28 after randomization
  thrombocytopenia (< 100 000 platelets/mm3)
Rate of thrombosis of a large venous axis (randomization stage) | Until ICU discharge or day 28 after randomization
  thrombosis of a large venous axis diagnosed by Doppler ultrasonography
Rate of hypophosphatemia (randomization stage) | Until ICU discharge or day 28 after randomization
  hypophosphatemia (defined as a serum phosphate concentration<0.6 mmol/l)
Rate of hyperkalemia (randomization stage) | Until ICU discharge or day 28 after randomization
  hyperkalemia (> 6.5 mmol/l)
Rate of hypernatremia (randomization stage) | Until ICU discharge or day 28 after randomization
  Hypernatremia (>150 mmol/l)
Rate of cardiac rhythm disorders (randomization stage) | Until ICU discharge or day 28 after randomization
  ventricular tachycardia, ventricular fibrillation, torsade de pointe or new episode of atrial fibrillation requiring medical treatment or external electric counter shock
Rate of pneumothorax (randomization stage) | Until ICU discharge or day 28 after randomization
Rate of hemothorax (randomization stage) | Until ICU discharge or day 28 after randomization
Rate of air embolism (randomization stage) | Until ICU discharge or day 28 after randomization
Number of arterio-venous fistulae (randomization stage) | Until ICU discharge or day 28 after randomization
Rate of pericarditis (randomization stage) | Until ICU discharge or day 28 after randomization
Rate of unexpected cardiac arrest (randomization stage) | Until ICU discharge or day 28 after randomization
Rate of hypothermia (randomization stage) | Until ICU discharge or day 28 after randomization
  Hypothermia (<34°C)
Percentage of patients receiving RRT at least once in the " delayed" RRT strategy arm (randomization stage) | Until ICU discharge or day 28 after randomization
Number of RRT sessions (randomization stage) | Until ICU discharge or day 28 after randomization
  Number of RRT sessions (until D28 after randomization) (analyzing alive or dead patients separately)
Time between randomization and RRT initiation (randomization stage) | Until ICU discharge or day 28 after randomization
Time to RRT weaning (randomization stage) | Until ICU discharge or day 28 after randomization
Time to renal function recovery (randomization stage) | Until ICU discharge or day 28 after randomization
Total cost of RRT-related consumables (randomization stage) | Until ICU discharge or day 28 after randomization
  catheters, solutions for RRT, membranes, and circuitry
Number of dialysis catheter-free day (randomization stage) | Until ICU discharge or day 28 after randomization
Rate of catheter-related bloodstream infection (randomization stage) | Until ICU discharge or day 28 after randomization
  both dialysis and non-dialysis catheters
Barthel ADL (activity of daily living) index (randomization stage) | Day 60 after randomization
  Barthel ADL index at D60 (an index of activities of daily living)
Percentage of patients with a decisions to withhold or withdraw life support therapies (randomization stage) | Until ICU discharge or day 28 after randomization
Duration of ICU stay (observational and randomization stage) | Limited to 60 days after randomization
Duration of hospital stay (observational and randomization stage) | Limited to 60 days after randomization
ICU mortality (observational and randomization stage) | Limited to 60 days after randomization
Day 28 mortality (observational and randomization stage) | Day 28 after inclusion
Day 60 mortality (observational and randomization stage) | Day 60 after inclusion
Hospital mortality (observational and randomization stage) | Limited to 60 days after randomization
Ventilator free-days (observational and randomization stage) | Day 28 after inclusion
RRT indications (observational and randomization stage) | Day 28 after inclusion
  Reason(s) to start RRT during observational stage will be assessed
RRT modalities (observational and randomization stage) | Day 28 after inclusion
  CRRT (continuous renal replacement therapy) , IHD (Intermittent Hemodialysis), other
Duration of RRT | Until ICU discharge or day 28 after randomization
Time to renal function recovery (observational and randomization stage) | Until ICU discharge or day 28 after randomization
  Renal function recovery will be defined by spontaneous diuresis >1000 ml/24h without diuretic administration or >2000 ml/24h, in patients receiving diuretics.
Time to spontaneous decrease in creatinine | Until ICU discharge or day 28 after randomization
  Spontaneous decrease of serum creatinine for 2 consecutive days without need for RRT during the following 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Didier DREYFUSS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (41):
- France (40):
  - CH Alès, Alès
  - CHU Amiens, Amiens
  - CH Avignon, Avignon
  - Groupe Hospitalier Carnelle-Portes de l'Oise Site Beaumont / Oise, Beaumont-sur-Oise
  - Hopital Nord Franche Comté - Belfort, Belfort
  - CH Béthune Beuvry - Germont et Gauthier, Béthune
  - CHU Avicenne - APHP, Bobigny
  - CHU Ambroise Paré - APHP, Boulogne-Billancourt
  - CH Bourg en Bresse / Fleyriat, Bourg-en-Bresse
  - Gabriel Montpied - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Louis Mourier - APHP, Colombes
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor - APHP, Créteil
  - CH Dieppe, Dieppe
  - Hôpital François Mitterand - CHU Dijon, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CH Dr Schaffner - Lens, Lens
  - Hôpital Roger Salengro / CHRU Lille, Lille
  - Centre Hospitalier Bretagne sud - Lorient, Lorient
  - GH Edouard Herriot - Lyon, Lyon
  - Hôpital Nord - Anesthésie Réa - APHM, Marseille
  - Hôpital Nord - DRIS - APHM, Marseille
  - La Timone - APHM, Marseille
  - Hopital de Mercy, CHR Metz-Thionville, Metz
  - Hôpital Lapeyronie - CHU Montpellier, Montpellier
  - Hôpital St Eloi - CHU Montpellier, Montpellier
  - Hotel Dieu - Anesthésie Réanimation - CHU Nantes, Nantes
  - Hotel Dieu - Réanimation MIR - CHU Nantes, Nantes
  - Hôpital Nord Laennec - CHU Nantes, Nantes
  - CHU Nimes - Caremeau, Nîmes
  - Chu Hegp - Aphp, Paris
  - CHU Pitiè Salpêtrière - Pneumologie et réanimation médicale - APHP, Paris
  - CHU Pitié-Salpêtrière - Réanimation médicale - APHP, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - CH René DUBOS, Pontoise
  - CHU Charles Nicolle, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CH André Mignot, Versailles
- CHU pointe à Pitre / Abymes, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Gaudry S, Hajage D, Martin-Lefevre L, Lebbah S, Louis G, Moschietto S, Titeca-Beauport D, Combe B, Pons B, de Prost N, Besset S, Combes A, Robine A, Beuzelin M, Badie J, Chevrel G, Bohe J, Coupez E, Chudeau N, Barbar S, Vinsonneau C, Forel JM, Thevenin D, Boulet E, Lakhal K, Aissaoui N, Grange S, Leone M, Lacave G, Nseir S, Poirson F, Mayaux J, Asehnoune K, Geri G, Klouche K, Thiery G, Argaud L, Rozec B, Cadoz C, Andreu P, Reignier J, Ricard JD, Quenot JP, Dreyfuss D. Comparison of two delayed strategies for renal replacement therapy initiation for severe acute kidney injury (AKIKI 2): a multicentre, open-label, randomised, controlled trial. Lancet. 2021 Apr 3;397(10281):1293-1300. doi: 10.1016/S0140-6736(21)00350-0. PMID 33812488
- [Derived] Meraz-Munoz AY, Bagshaw SM, Wald R. Timing of kidney replacement therapy initiation in acute kidney injury. Curr Opin Nephrol Hypertens. 2021 May 1;30(3):332-338. doi: 10.1097/MNH.0000000000000707. PMID 33767061
- [Derived] Gaudry S, Hajage D, Martin-Lefevre L, Louis G, Moschietto S, Titeca-Beauport D, La Combe B, Pons B, de Prost N, Besset S, Combes A, Robine A, Beuzelin M, Badie J, Chevrel G, Reignier J, Bohe J, Coupez E, Chudeau N, Barbar S, Vinsonneau C, Forel JM, Thevenin D, Boulet E, Lakhal K, Aissaoui N, Grange S, Leone M, Lacave G, Nseir S, Poirson F, Mayaux J, Asehnoune K, Geri G, Klouche K, Thiery G, Argaud L, Ricard JD, Quenot JP, Dreyfuss D. The Artificial Kidney Initiation in Kidney Injury 2 (AKIKI2): study protocol for a randomized controlled trial. Trials. 2019 Dec 16;20(1):726. doi: 10.1186/s13063-019-3774-9. PMID 31843007